CLINICAL TRIAL: NCT03766412
Title: High School Start Time and Adolescent Migraine Frequency
Brief Title: High School Start Time and Teen Migraine Frequency
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: High School Start Time Study
Record Dates: First submitted 2018-10-11; First posted 2018-12-06 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2018-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- School start time 8:30 AM or later: These are high schoolers with migraine who attend a school that begins at 8:30 AM or later (i.e. follows AAP recommendation re: high school start time).
  Interventions: Other: High School start time
- School start time earlier than 8:30: These are high schoolers with migraine who attend a school that begins earlier than 8:30 AM (i.e. does not follow AAP recommendation re: high school start time).
  Interventions: Other: High School start time

INTERVENTIONS:
Other: High School start time — The time that the school starts

SUMMARY:
Migraine is common in adolescents and can cause missed school and disability.

The American Academy of Pediatrics (AAP) recommends that high schools start no earlier than 8:30 AM in order to accommodate the physiologic needs of adolescents-whose brains naturally want to fall asleep later and wake up later and who still need to get at least 8 hours of sleep per night to function optimally-however, only about 18% of US high schools comply with this AAP recommendation. There is a relationship between adequate sleep and migraine. The investigators aim to determine whether high school students with migraine who attend high schools that comply with this AAP recommendation have lower migraine frequency than those that do not.

If so, it would argue for advocating for changes in high school policy to optimize health of adolescents with migraine.

DETAILED DESCRIPTION:
Study design: This is an observational study of high-school students in the U.S. who have migraine and who attend a standard high school (i.e. are not home schooled or online schooled). They will complete a one-time online survey answering questions about their headaches and their schedule--particularly schedule aspects related to school and sleep.

ELIGIBILITY:
Inclusion criteria:

1. Live in the U.S.
2. In 9th-12th grade
3. Attends a high school that is outside of the home (i.e. not home-schooled or online schooled)
4. High school has a consistent start time all 5 days of the week
5. Has migraine by International Classification of Headache Disorders criteria
6. Can read and write in English

Exclusion criteria: NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: U.S. High school students with migraine
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Headache days per month | Last 30 days
  How many headache days experienced in the last month

SECONDARY OUTCOMES:
Hours of sleep on typical school night | Last 30 days
  Respondent's estimate of hours of sleep on a typical school night
Typical bedtime on school night | Last 30 days
  Respondent's estimate of typical bedtime on school night
Typical wake up time on a school day | Last 30 days
  Respondent's estimate of typical wakeup time on a school day
Number of missed breakfasts in a typical school week | Last 30 days
  Respondent's estimate of how many times they miss breakfast in a typical school week
Acute headache medication days per month | Last 30 days
  How many days per month respondent uses acute headache medication
PedMIDAS (Pediatric Migraine Disability Assessment Scale) | Last 90 days
  Headache related disability score--Total score ranges from 0-246

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Gelfand, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gelfand AA, Pavitt S, Greene K, Szperka CL, Irwin S, Grimes B, Allen IE. High School Start Time and Migraine Frequency in High School Students. Headache. 2019 Jul;59(7):1024-1031. doi: 10.1111/head.13535. Epub 2019 Apr 24. PMID 31016722